CLINICAL TRIAL: NCT00333632
Title: Restorative Sleep: Effect of Dexmedetomidine
Brief Title: Effect of Dexmedetomidine Upon Sleep Postoperatively
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00007964; 8306 (Other: Duke legacy protocol number)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2011-06

CONDITIONS: Sleep
Keywords: Sleep; Dexmedetomidine; Postoperative care; Sedation
MeSH Terms: interventions — Dexmedetomidine; Propofol; Midazolam; Fentanyl; Isoflurane

INTERVENTIONS:
Drug: Dexmedetomidine
Drug: Propofol
Drug: Midazolam
Drug: Fentanyl
Drug: Isoflurane

SUMMARY:
The purpose of this study is to determine whether an intravenous infusion of dexmedetomidine administered to surgical patients intra-operatively will improve the characteristics of sleep post-operatively.

DETAILED DESCRIPTION:
Physiological similarities exist between the anesthetized state and sleep. Pathways within the brain controlling sleep and wakefulness are also affected by anesthesia. One significant difference between the states of anesthesia and sleep is the ability to respond whenever a relatively mild stimulus is applied, e.g. verbal command or gently shaking. Interestingly, this feature of arousability is seen when dexmedetomidine is used for sedation but is absent when alternative intravenous anesthetic agents, e.g. propofol, are used to provide similar degree of sedation. Recent studies have shown that dexmedetomidine acts on receptors located within the locus ceruleus, which are responsible for both sleep and anesthesia.

During a recent study volunteers received an infusion of dexmedetomidine during the afternoon prior to remaining under study conditions for the duration of the night. The study was not designed to measure sleep but anecdotal reporting from the participants suggested that they were able to resume their normal day's activities whilst the subject receiving placebo felt extremely fatigued from lack of sleep. This prompted the establishment of a pilot study to determine if dexmedetomidine could provide restorative sleep to people under disturbed sleep conditions i.e. postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo elective lower extremity orthopaedic surgery (free vascular fibular graft)
* ASA 1 or 2
* Body Mass Index 20 - 30
* Procedure to be done under combined epidural and general anesthesia

Exclusion Criteria:

* Sleep disturbance
* Insomnia
* Sleep apnea
* Female (pregnant)
* Contra-indication to placement of epidural anesthesia

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Measurements of sleep quality during postoperative period:Epworth Sleepiness Scale
Completion of sleep log
Subjects will also be asked to complete Visual Analogue Scales (VAS) of sleep and daytime sleepiness.

SECONDARY OUTCOMES:
The quality of postoperative recovery (QoR) and the presence of fatigue (Brief Fatigue Inventory)
Subjects will also be asked to complete Visual Analogue Scale (VAS) of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States